CLINICAL TRIAL: NCT07157566
Title: Effects of Mindfulness Practice and E-health Information Push on E-health Literacy, Media Literacy, Food Literacy, and Mindfulness Skills Among University Students in Macau
Brief Title: From Health Information to Health Decisions Integrating Mindfulness Into Digital Learning and Daily Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Macau (Other)
Responsible Party: Principal Investigator, Siman Lei, Assistant Professor, University of Macau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HE-0947-2025
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Health Literacy; Food Literacy; Media Literacy; E-health Literacy
Keywords: Randomized Controlled Trial; Health literacy; Media literacy; Food Literacy; Mindfulness; Critical thinking; Decision making; e-health literacy
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness Group (Experimental): Participants in this group will engage in an 8-week program integrating mindful eating and mindful movement practices into their regular physical education classes. Each session includes 10 minutes of mindful eating exercises designed to enhance awareness of hunger and satiety cues, sensory experiences of food, and emotional responses to eating. The final 10 minutes of each session consist of mindful movement exercises, combining physical postures and movements with mindfulness techniques to improve food literacy, physical literacy, and social-emotional competencies.
  Interventions: Behavioral: Mindfulness
- E-health Group (Experimental): Participants in this group will receive two digital health information materials per week via Moodle or email, each requiring approximately 5-10 minutes of reading time. The topics of the materials include: health literacy; nutrition; exercise and stress; mental health and sleep; and behavior change and integration. These aim to enhance participants' digital health literacy, media literacy, and related competencies.
  Interventions: Behavioral: e-Health Literacy
- Mindfulness + E-health Group (Experimental): Participants in this group will engage in an 8-week program that integrates mindful eating and mindful movement practices into their regular physical education classes, while also receiving digital health information materials to enhance their e-health literacy. The program is designed to improve participants' food literacy, physical literacy, social-emotional competencies, e-health literacy, and media literacy through a combination of practical exercises and educational content.
  Interventions: Behavioral: Mindfulness; Behavioral: e-Health Literacy
- Control Group (No Intervention): Participants in this group will follow their regular physical education classes without incorporating any mindfulness practices or digital health information materials. The control group will engage in standard activities and curricula designed for university physical education, which may include various physical training, sports, and theoretical instruction related to health and fitness.

INTERVENTIONS:
Behavioral: Mindfulness — Structured over 8 weeks (twice weekly) with dual modules (dietary + movement), this group employs Mindfulness-Based Eating Awareness Training (MB-EAT) to improve mind-body awareness. Week 1 establishes foundational practices through mindful eating concepts and introductory yoga; Weeks 2-4 systematically train awareness of hunger/satiety cues using partner breathing techniques, postural alignment, and group-assisted stretching; Week 5 analyzes emotional eating triggers while integrating therapeutic yoga for emotional regulation; Weeks 6-7 foster body acceptance and autonomous food choices; the program concludes with closing rituals. Rooted in Mindfulness-Based Stress Reduction (MBSR), it strengthens interoceptive awareness, non-judgmental self-acceptance, and emotional management to transform dysfunctional eating patterns.
  Arms: Mindfulness + E-health Group; Mindfulness Group
Behavioral: e-Health Literacy — This 8-week program (twice weekly) aims to enhance participants' ability to access, evaluate, and apply digital health information. It progresses through sequential modules: Week 1 introduces e-Health literacy fundamentals and physical activity principles; Weeks 2-3 focus on nutritional assessment and personalized planning; Week 4 addresses sleep health; Weeks 5-7 train health information retrieval skills, including database navigation and source reliability verification; the final week hones critical appraisal capabilities. The intervention is based on the e-Health Literacy 3.0 model and cultivates three core competencies: digital navigation, information discernment, and evidence-based decision-making, enabling participants to independently navigate the digital health ecosystem.
  Arms: E-health Group; Mindfulness + E-health Group

SUMMARY:
This research project aims to explore how combining e-health literacy with mindfulness practices can help university students navigate the complex landscape of e-health information and make more informed, healthier choices. Specifically, the study will assess the current levels of e-health literacy, food literacy, and media literacy among university students, and examine how these factors are related to critical thinking, decision-making confidence, and overall well-being. The project will involve a 4-arm design, including: (1) a mindfulness group, (2) an e-health group, (3) a mindfulness + e-health Group, and (4) a Control Group. Participants in the intervention groups will engage in short mindfulness exercises focused on mindful eating and movement during break times and cool-down sessions of their Physical Education (PE) classes. Additionally, digital health content (e.g., videos and articles) will be provided to enhance e-health literacy. This could lead to better-informed, more confident students who are able to make healthier choices in their daily lives, both during their university years and into the future.

Study Aim

To evaluate the effectiveness of an 8-week intervention delivered during PE classes, comparing the effects of:

1. Mindfulness Group 2. E-health Group 3. Mindfulness + E-health Group 4. Control Group The intervention will assess changes in students' e-health literacy, food literacy, media literacy, critical thinking, self-compassion and decision-making self-efficacy over time, with assessments at pre-test, post-test, and 4-week follow-up.

Study Hypotheses:

1. Students in the mindfulness group, e-health group, and combined group will show significantly greater improvements in all outcome measures from pre-test to post-test compared to the control group.
2. The combined group will demonstrate the greatest gains in literacy and cognitive outcomes, due to the additive effect of both interventions.
3. Improvements will be maintained at the 4-week follow-up, particularly in the combined group.

DETAILED DESCRIPTION:
This study aims to explore the effects of mindfulness practice and e-health interventions on e-health literacy, media literacy, food literacy, critical thinking, and decision-making abilities among university students.

Research Objectives: To investigate the impact of mindfulness practice and e-health interventions on university students' e-health literacy, media literacy, food literacy, critical thinking, and decision-making abilities, and to evaluate their short-term effectiveness.

Participants: 268 university students aged between 18 and 25 who are willing to participate in mindfulness activities during and after class and receive e-health-related information.

Study Procedure:

1. Baseline Assessment: Includes questionnaires on e-health literacy, media literacy, critical thinking, and food literacy, as well as tests conducted using E-Prime software.
2. Intervention: Participants will take part in an 8-week program during their physical education classes and leisure time. They will be randomly assigned to one of four groups:

   Mindfulness Group: Engage in mindful eating and mindful movement exercises during each physical education class (approximately 20 minutes).

   E-health Group: Read or listen to two push notifications of e-health information per week, covering topics such as health management, stress and sleep, nutrition, and behavior change.

   Combined Group: Participate in both mindfulness practice and receive e-health information.

   Control Group: Receive no additional intervention and participate only in regular physical education classes.
3. Post-Intervention Assessment: Immediately after the 8-week intervention, participants will complete the same questionnaires and E-Prime tests as at baseline to assess immediate effects.
4. Follow-Up Assessment: Four weeks after the intervention ends, the same set of measurements will be conducted again to evaluate the sustainability of the intervention effects.
5. Interviews (Optional): With your consent, semi-structured or unstructured interviews may be conducted during and after the intervention to gain in-depth insights into your experiences and perceptions.

Statistical Analysis: A mixed-design analysis of variance (ANOVA) or analysis of covariance (ANCOVA) will be used to compare the effects across different time points. Post-hoc tests will be conducted to identify specific differences between the various groups and across different time points. The significance level will be set at a p-value of less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

Mindfulness Group

1. Currently enrolled in a Physical Education (PE) class.
2. Aged between 18 and 25 years.
3. Willing to participate in the 8-week intervention and provide informed consent.
4. Generally healthy and able to engage in physical activity.
5. Proficient in Chinese.

E-health Group

1. Currently enrolled in a Physical Education (PE) class.
2. Aged between 18 and 25 years.
3. Willing to participate in the 8-week intervention and provide informed consent.
4. Generally healthy and able to engage in physical activity.
5. Proficient in Chinese.

Mindfulness + E-health Group

1. Currently enrolled in a Physical Education (PE) class.
2. Aged between 18 and 25 years.
3. Willing to participate in the 8-week intervention and provide informed consent.
4. Generally healthy and able to engage in physical activity.
5. Proficient in Chinese.

Control Group

1. Currently enrolled in a Physical Education (PE) class.
2. Aged between 18 and 25 years.
3. Willing to participate in the 8-week intervention and provide informed consent.
4. Generally healthy and able to engage in physical activity.
5. Proficient in Chinese.

Exclusion Criteria:

Mindfulness Group

1. Currently studying in medical, nutrition, or health-related fields.
2. Pregnant or lactating.
3. Severe mental health conditions or cognitive impairments affecting participation.
4. Currently participating in other mindfulness or digital health programs.
5. Involved in competitive sports (e.g., varsity athletes).
6. Recent major life events (e.g., trauma or major illness) within the last 6 months.
7. Unable to participate in PE classes due to medical or personal reasons.

E-health Group

1. Currently studying in medical, nutrition, or health-related fields.
2. Pregnant or lactating.
3. Severe mental health conditions or cognitive impairments affecting participation.
4. Currently participating in other mindfulness or digital health programs.
5. Involved in competitive sports (e.g., varsity athletes).
6. Recent major life events (e.g., trauma or major illness) within the last 6 months.
7. Unable to participate in PE classes due to medical or personal reasons.

Mindfulness + E-health Group

1. Currently studying in medical, nutrition, or health-related fields.
2. Pregnant or lactating.
3. Severe mental health conditions or cognitive impairments affecting participation.
4. Currently participating in other mindfulness or digital health programs.
5. Involved in competitive sports (e.g., varsity athletes).
6. Recent major life events (e.g., trauma or major illness) within the last 6 months.
7. Unable to participate in PE classes due to medical or personal reasons.

Control Group

1. Currently studying in medical, nutrition, or health-related fields.
2. Pregnant or lactating.
3. Severe mental health conditions or cognitive impairments affecting participation.
4. Currently participating in other mindfulness or digital health programs.
5. Involved in competitive sports (e.g., varsity athletes).
6. Recent major life events (e.g., trauma or major illness) within the last 6 months.
7. Unable to participate in PE classes due to medical or personal reasons.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 268 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
eHealth Literacy Scale (eHEALS) | From enrollment to the end of intervention at 8 weeks, and a 4-week follow up
  This scale is designed to assess an individual's perceived comprehensive ability to use information technology to solve health-related problems, which includes skills such as searching for, evaluating, and applying online health information. Based on the e-Health Literacy Model, the scale covers six core competencies: traditional literacy, health literacy, information literacy, scientific literacy, media literacy, and computer literacy. The scale consists of 8 core items, from question 3 to question 10, each rated on a 5-point Likert scale ranging from 1 = strongly disagree to 5 = strongly agree. The total score is calculated only for the core items, with a possible range of 8 to 40 points. The scale demonstrates high internal consistency reliability, with a Cronbach's α of 0.88. The unidimensional structure is stable, with principal component analysis explaining 56% of the variance and factor loadings ranging from 0.60 to 0.84.
Media Health Literacy Scale (MeHLit) | From enrollment to the end of intervention at 8 weeks, and a 4-week follow up
  This scale is designed to assess adults' abilities to interpret health-related information in the media. Its design is based on an integrated framework combining health literacy and media literacy. The final version of the scale consists of 21 items, divided into five dimensions: Goal Appraisal Skills, Content Appraisal Skills, Implied Meaning Appraisal Skills, Visual Comprehension Skills, and Audience Appraisal Skills. Scoring is conducted using a 5-point Likert scale: Never (0 points) to Always (4 points). The total score is the sum of all item scores, ranging from 0 to 84 points. The scale demonstrates excellent content validity, with a Content Validity Index (CVI) of 0.93 and a Content Validity Ratio (CVR) of 0.87. Exploratory Factor Analysis extracted a 5-factor structure that explains 60.25% of the total variance. Confirmatory Factor Analysis indicated a good model fit (RMSEA = 0.051, CFI = 0.93). The overall scale's Cronbach's α is 0.91.
Food Literacy Evaluation Questionnaire (Chinese version, FLEQ-Ch) | From enrollment to the end of intervention at 8 weeks, and a 4-week follow up
  This scale is designed to assess the food literacy of Chinese residents. The questionnaire was adapted from the original FLEQ (Food Literacy Evaluation Questionnaire) and consists of 15 items divided into three main dimensions: Planning and Management, Selection, and Preparation.
  The "Planning and Management" dimension includes 7 items evaluating participants' ability to plan meals in advance, create shopping lists, include all food groups in meals, consider healthy choices, manage funds for purchasing healthy foods, and learn ways to access healthy foods. Scoring ranges from 0 (Never) to 3 (Always). The total score ranges from 0 to 45, with higher scores indicating higher levels of food literacy.
  The FLEQ-Ch demonstrates good psychometric properties, with internal consistency ranging from 0.869 to 0.955 and test-retest reliability coefficients ranging from 0.941 to 0.952.
Assessment Tools for Critical Thinking and Decision-Making Abilities | From enrollment to the end of intervention at 8 weeks, and a 4-week follow up
  The tasks used in this study to assess critical thinking and decision-making abilities were executed using E-Prime 3.0 software (Psychology Software Tools, Inc.) for stimulus presentation and response data collection. E-Prime is widely used in psychological and behavioral research, with its key advantage being the ability to control the presentation timing and duration of visual and auditory stimuli with millisecond precision, while simultaneously recording participants' response times and accuracy rates. It shows potential for application in measuring critical thinking and decision-making abilities in the health domain. These two abilities are crucial for effective personal health management.
  Although E-Prime is not specifically designed to measure critical thinking and decision-making skills, its functionality is more oriented toward executing experimental tasks. It can indirectly assess cognitive processes related to these abilities.

SECONDARY OUTCOMES:
New Media Literacy Scale (NMLS) | From enrollment to the end of intervention at 8 weeks, and a 4-week follow up
  This scale aims to comprehensively assess college students' new media literacy in the digital era. It is specifically divided into four dimensions: Functional Consumption, Critical Consumption, Functional Prosumption, and Critical Prosumption. The scale consists of 35 items and employs a 5-point Likert scale scoring system, ranging from 1 = strongly disagree to 5 = strongly agree. During scoring, the four dimensions are independently summed as follows: Functional Consumption (FC, 7-35 points), Critical Consumption (CC, 16-55 points), Functional Prosumption (FP, 7-35 points), and Critical Prosumption (CP, 10-50 points). Alternatively, all items can be summed to obtain an overall score (35-175 points). The Cronbach's α for each dimension ranges from 0.85 to 0.93, while the overall scale α = 0.95. All item-total correlations are >0.30, and the inter-dimensional correlations are moderate (r = 0.44-0.63).
Self-compassion short form (SCS-SF) | From enrollment to the end of intervention at 8 weeks, and a 4-week follow up
  The scale retains the original six-dimensional structure: Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness, and Over-Identification. It also supports a higher-order single-factor model for "overall self-compassion." The total score of the scale demonstrates high internal consistency reliability, with Cronbach's α ≥ 0.86, and shows an extremely high correlation with the total score of the full version (r ≥ 0.97).
  For scoring, items in the Self-Judgment (SJ), Isolation (I), and Over-Identification (OI) dimensions must be reverse-scored (e.g., an original score of 5 is converted to 1). The scores of the six subscales are then summed (each subscale consists of 2 items, e.g., the SK subscale = Item 2 + Item 6). The total score ranges from 12 to 60 points, with higher scores indicating greater levels of self-compassion.
Decision Self-Efficacy Scale | From enrollment to the end of intervention at 8 weeks, and a 4-week follow up
  This scale was developed by A.M. O'Connor in 1995 to measure an individual's confidence in their own decision-making abilities and their self-efficacy in making informed choices. The scale consists of 11 uniform items covering four core competencies: obtaining information; understanding and application; communication and expression; and autonomous decision-making. This study uses a 5-point version of the scale. The scoring method involves three steps: (1) sum the scores of the 11 items, (2) divide the total by 11, and (3) multiply by 25 to obtain a standardized score ranging from 0 to 100. (where 0 represents "very low self-efficacy" and 100 represents "very high self-efficacy") Psychometric properties indicate that the 5-point Likert version achieved a Cronbach's α of 0.92.
Decisional Conflict Scale | From enrollment to the end of intervention at 8 weeks, and a 4-week follow up
  The scale is a standardized instrument developed by A.M. O'Connor to measure an individual's level of decisional conflict when facing choices. Its definition encompasses three main domains: (1) uncertainty in choosing options; (2) modifiable factors that exacerbate uncertainty; and (3) decision effectiveness. The study used the traditional statement format version, which consists of 16 items. It employs a 5-point Likert scoring system, with response options ranging from "0 = strongly disagree" to "4 = strongly agree." Scoring is performed by assigning values to the response options, calculating the average score for subscales or the total score, and then multiplying by 25. The subscales are: Informed; Values Clarity; Support; Uncertainty; and Effective Decision. The scale demonstrated excellent psychometric properties, with a Cronbach's α > 0.78, high test-retest reliability, and the ability to discriminate between deciders and delayers (effect size 0.4-0.8).
Five Facet Mindfulness Questionnaire (FFMQ-C-SF) | From enrollment to the end of intervention at 8 weeks, and a 4-week follow up
  This questionnaire is a reliable and valid mindfulness measurement tool designed for Chinese populations. Its origins can be traced back to the English version of the Five Facet Mindfulness Questionnaire (FFMQ), which was translated and simplified to form a 20-item short form covering five dimensions: Describing, Acting with Awareness, Observing, Nonjudging, and Nonreactivity.
  Scoring is conducted using a 5-point Likert scale, with responses ranging from "1 = Never or very rarely true" to "5 = Very often or always true." The scores of the five dimensions are then summed, yielding a total score ranging from 20 to 100.
  The scale demonstrates good internal consistency (Cronbach's alpha = 0.77) and high correlation (r = 0.96 with the full FFMQ-C), making it an ideal choice for assessing mindfulness in both clinical and research setting.
International Fitness Scale (IFIS) | From enrollment to the end of intervention at 8 weeks, and a 4-week follow up
  This study utilized the International Fitness Scale (IFIS) for physical fitness assessment. The scale employs a 5-point Likert scale, with scoring ranging from "1 = Very poor" to "5 = Very good." The IFIS comprises five components: overall physical fitness, cardiorespiratory endurance, muscular strength, speed and agility, and flexibility.
  The scale has been reported to demonstrate acceptable validity and reliability in young populations. A total of 276 participants aged 18-30 were recruited for a reliability study. The results indicated that the IFIS exhibits acceptable reliability in young adults, with an average Kappa value of 0.59. Kappa values ranging from 0.54 to 0.65 are considered to indicate "moderate" to "good" reliability.
Critical Thinking Self-assessment Scale (CTSAS) | From enrollment to the end of intervention at 8 weeks, and a 4-week follow up
  The CTSAS (Critical Thinking Self-Assessment Scale) is a self-assessment tool developed based on Facione's six-dimensional model of critical thinking. It is designed to evaluate the critical thinking abilities of higher education students. This study employs a simplified version consisting of 60 items. The distribution of items is as follows: Interpretation (9 items), Analysis (11 items), Evaluation (7 items), Inference (13 items), Explanation (10 items), and Self-regulation (10 items). The scale uses a 7-point Likert scoring system, ranging from 0=Never to 6=Always. Users can calculate sub-scores for each dimension or a total overall score. Higher scores indicate stronger critical thinking skills. This simplified version has demonstrated excellent reliability and validity. The overall scale's Cronbach's α reached 0.969, and the α values for the individual dimensions ranged from 0.772 to 0.905.

CONTACTS AND LOCATIONS:
Overall Officials: SiMan LEI, Doctoral, Principal Investigator — University of Macau
Locations (2):
- Macau (2):
  - UM Sports Complex (N8) , Avenida da Universidade Taipa, Macau, China, Macao
  - University of Macau, Macao

IPD SHARING:
Plan to Share IPD: No